CLINICAL TRIAL: NCT06260631
Title: Efficacy of High-intensity Laser Acupuncture in Patients With Chronic Non-specific Low Back Pain: a Double-blinded, Randomized Controlled Trial
Brief Title: Efficacy of High-intensity Laser Acupuncture in Patients With Chronic, Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: King Khalid University (Other)
Responsible Party: Principal Investigator, Doaa Ayoub Elimy Mohammed, Lecturer of physical therapy for basic science department., faculty of physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004807
Record Dates: First submitted 2024-02-05; First posted 2024-02-15 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Chronic Nonspecific Low-back Pain
Keywords: low back pain; high-intensity laser acupuncture; peak torque; power; functional disability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: high-intensity laser acupuncture and exercise therapy program
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity laser acupuncture and an exercise therapy program. (Experimental): The patients will receive high-intensity laser acupuncture and an exercise therapy program.three times a week for four weeks.
  Interventions: Device: high-intensity laser acupuncture and Exercise therapy program
- sham laser acupuncture and an exercise therapy program. (Sham Comparator): The patients will receive a sham acupuncture laser and an exercise therapy program three times a week for four weeks.
  Interventions: Other: Sham laser acupuncture

INTERVENTIONS:
Device: high-intensity laser acupuncture and Exercise therapy program — The experimental group will receive high-intensity lasers and the treatment will be performed at 15 acupuncture points: unilateral GV3, GV4, and GV5, and bilateral BL 20, BL23, BL24, BL25, BL40 and GB30.
  Exercise therapy program
  The patients will perform an exercise therapy program in the form of:
  * strengthening exercises for abdominal and back muscles,
  * lumbar stabilization exercises.
  * stretching exercises.
  Other Names: high-power laser acupuncture
  Arms: high-intensity laser acupuncture and an exercise therapy program.
Other: Sham laser acupuncture — Sham laser acupuncture and exercise therapy program
  The patients will receive a sham laser.acupuncture and an exercise therapy program in the form of:
  * strengthening exercises for abdominal and back muscles,
  * lumbar stabilization exercises.
  * stretching exercises.
  Arms: sham laser acupuncture and an exercise therapy program.

SUMMARY:
The purpose of this study is to investigate the efficacy of high-intensity laser acupuncture on peak torque, power of trunk extensors and flexors, back pain, range of motion, function, and satisfaction in patients with chronic nonspecific low back pain (CNLBP).

DETAILED DESCRIPTION:
Chronic nonspecific low back pain (CNLBP) is a persistent back pain that affects people of all ages and contributes to the global disease burden. Treatment focuses on reducing pain and its consequences. High-intensity laser therapy is a non-invasive, painless modality that can be easily administered for various conditions. It has been proven to significantly reduce pain, with anti-inflammatory, anti-edematous, and analgesic effects. Laser photobiomodulation (PBM) therapy is a non-invasive and painless method that stimulates cells, pain receptors, and the immune system and can cause vasodilation and analgesic effects. Acupuncture is a common complementary therapy that has been proven to treat musculoskeletal pain and enhance muscle strength, and high-intensity laser acupuncture (HILA) has been promoted as an alternative to traditional needle acupuncture. HILA, as a non-invasive treatment, combines the efficacy of high-intensity laser and acupuncture in musculoskeletal pain management. Due to a lack of research, this study will examine the effects of HILA on peak torque and power of the trunk extensors and flexors, back pain, range of motion, function, and satisfaction in patients with chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. The patients had CNSLBP with age from 20 to 40 years from both genders.
2. Patients will be referred from an orthopedist with diagnosis of chronic low back pain without underlying pathological causes.
3. The patients with chronic nonspecific low back pain more than 3months. Minimum pain intensity of 30 mm on the visual analogue scale (VAS) for pain, which ranges from 0 to 100 mm.
4. Patients with normal BMI ranges between 18.5:24.9 kg/m2.
5. The study populations must be willing to participate in the study

Exclusion Criteria:

1. Neurological, infectious diseases and systemic illness such as rheumatologic diseases,systemic lupus erythematosus, diabetes mellitus type I or II.
2. Psychiatric/mental deficit.
3. Patients who had a previous surgical history (within 6 months) will also excluded.
4. participation in other treatment within the previous 3 month.
5. Pregnancy.
6. History of spinal fracture, tumor, osteoporosis
7. use of medication, such as corticosteroids, anticonvulsants, and anti-inflammatory drugs that may affect the outcome of the study.
8. prior history of adverse effects to physical stimulation therapy.
9. significant physical or mental deficiencies preventing a clear understanding of the study procedure.
10. spinal stenosis, thyroid dysfunctions, obesity, pace-maker.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
peak torque | up to four weeks
  Isokinetic dynamometer will be used for measuring peak torque of back extensors and flexors.
peak torque | follow up after 1 month
  Isokinetic dynamometer will be used for measuring peak torque of back extensors and flexors..
Average Power | up to four weeks
  Isokinetic dynamometer will be used for measuring Average Power in watts for both back extensors and flexors.
Average Power | follow up after 1 month
  Isokinetic dynamometer will be used for measuring Average Power in watts for both back extensors and flexors.

SECONDARY OUTCOMES:
Pain Intensity | up to four weeks
  Visual Analogue Scale (VAS) will be used by the patient to mark his/her level of pain between 0 to100 milliliters line. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Pain Intensity | follow up after 1 month
  Visual Analogue Scale (VAS) will be used by the patient to mark his/her level of pain between 0 to100 milliliters line. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
lumbar flexion and extension ROM assessment | up to four weeks
  Modified-modified Schober test will be used to assess ROM of lumbar flexion and extension
lumbar flexion and extension ROM assessment | follow up after 1 month
  Modified-modified Schober test will be used to assess ROM of lumbar flexion and extension
Disability | up to four weeks
  Arabic version of Oswestry Disability Index (ODI) will be used for assessment of functional disability.
Disability | follow up after 1 month
  Arabic version of Oswestry Disability Index (ODI) will be used for assessment of functional disability.
patient Satisfaction | up to four weeks
  The satisfaction VAS will be used to measure patient satisfaction. The patient will be by placing an indicator at 0 to100 milliliters line. Zero usually represents 'no satisfaction at all' whereas the upper limit represents 'the best satisfaction ever'.
patient Satisfaction | follow up after 1 month
  The satisfaction VAS will be used to measure patient satisfaction. The patient will be by placing an indicator at 0 to100 milliliters line. Zero usually represents 'no satisfaction at all' whereas the upper limit represents 'the best satisfaction ever'.

CONTACTS AND LOCATIONS:
Locations (1):
- Doaa Ayoub Elimy, Giza, Egypt